CLINICAL TRIAL: NCT06233890
Title: The Analysis of Fatigue on Tyrosine Kinase Inhibitor Therapy in Chronic Myeloid Leukaemia
Acronym: TIRE
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22HH7973
Record Dates: First submitted 2024-01-08; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Chronic Myeloid Leukemia; Chronic Myeloid Leukemia, Chronic Phase; Fatigue; Sleep Disturbance
Keywords: Tyrosine kinase inhibitor; chronic myeloid leukaemia; sleep disturbance; fatigue; Activin B; L-carnitine
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase; Fatigue; Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fatigue: Group 1: Fatigue present for more than 6 months with impairment in daily life activities.
  Fatigue will be assessed using two validated fatigue questionnaires completed at the screening visit. The Chalder fatigue scale (CFQ) is an 11 item scale which assesses the severity of fatigue over the last 90 days and the Modified Fatigue Impact scale (MFIS), commonly used to determine the impact of fatigue on quality of life, assesses fatigue over the previous 30 days. Both scales are diagnostic tools in chronic disease associated fatigue. Scores on these scales will determine if patients are eligible. For this group a score > or = 5 for Chalder score and > or = 43 for the MFIS score.
  Interventions: Device: Motion watch
- Non -Fatigue: Group 2: no significant symptoms of fatigue on TKI therapy. Fatigue will be assessed using two validated fatigue questionnaires completed at the screening visit. The Chalder fatigue scale (CFQ) is an 11 item scale which assesses the severity of fatigue over the last 90 days and the Modified Fatigue Impact scale (MFIS), commonly used to determine the impact of fatigue on quality of life, assesses fatigue over the previous 30 days. Both scales are diagnostic tools in chronic disease associated fatigue. Scores on these scales will determine if patients are eligible. For this group a score < or = 2 for Chalder score and < or = 33 for the MFIS score.
  Interventions: Device: Motion watch

INTERVENTIONS:
Device: Motion watch — Actigraphy watch to be worn for 14 days

SUMMARY:
The goal of this clinical study is to gain essential insights into the relationship between Tyrosine kinase inhibitor (TKI) therapy and profound fatigue and abnormal sleep patterns using rest-activity monitoring (actigraphy) and peripheral blood biomarkers in patients with Chronic myeloid leukaemia in chronic phase. The main aims are to

1. Determine the variance of subjective and objective sleep disturbance
2. Determine the difference in serum biomarkers (activin B and L-carnitine)
3. Determine how thes findings concord/discord between treatment and control groups.

Participants will asked to undergo 2 weeks of actigraphy monitoring and keep a sleep diary during this time. Blood and urine samples will be taken for analysis.

Researchers will compare two groups (patients with fatigue and those without) to assess the differences between groups.

DETAILED DESCRIPTION:
The therapeutic landscape of CML has evolved significantly, as a result of targeted TKI therapy, over the past 2 decades with patients now experiencing a near normal life expectancy due to achievement of deep molecular responses. As a consequence, the appropriate management of drug related adverse events to ensure minimal impact on quality of life has never been more vital. Fatigue and sleep disturbance are commonly described and whilst it is evident that there is a strong correlation between fatigue and TKI therapy, the mechanism which drives this remains unknown. In general, the prevalence of TKI induced fatigue and predicting factors is largely unexplored. This exploratory, pilot study aims to examine the rest-activity patterns, blood parameters and fatigue related serum biomarkers of CML patients affected by fatigue on TKI therapy, and aims to provide insight into the association between fatigue and sleep disturbance on treatment. The pilot study aims to recruit 25 patients with profound fatigue on TKI therapy, for a minimum of 6 months with an impact on their activities of daily living. Additionally, we will recruit 25 further patients (age, gender and TKI matched) as a control cohort, who also have a diagnosis of Chronic Phase CML with no symptoms of fatigue. Validated fatigue questionnaires will be used (Chalder fatigue scale and the Fisk fatigue impact scale), these are key diagnostic tools in Fatigue associated disorders. TKI- fatigue syndrome (TKI-FS) symptoms can emulate the clinical pattern of Chronic Fatigue Syndrome (CFS) and this project would delineate congruence between CFS and TKI-FS. The patient cohort will also undergo actigraphy, this will be used in this study as a validated objective sleep measure, this method uses sophisticated analysis of movement to infer sleep/wake patterns. Actigraphy is non-invasive and can be used for several weeks, alongside a daily sleep diary, allowing collection of naturalistic sleep data as a participant goes about their normal activities. In addition, serum biomarkers such as activin B is a member of the activin family of proteins, which belongs to the TGF-β superfamily of growth and differentiation factors; activin B has been shown to be a potential serum biomarker in fatigue related disorders. In addition, L-carnitine is a vital molecular component in many metabolic pathways, the majority of the total body carnitine is located within skeletal muscle. Impairments in L-carnitine synthesis, transport or metabolism can result in primary or secondary deficiencies, which ultimately results in muscle weakness and fatigue. Assessment of both of these serum biomarkers in both the fatigue and control cohort may shed insight on whether there are significant differences between those patients with TKI-FS and the control group.

The aim of the study is to use the above stated modalities in order to gain further insight into the association between fatigue and sleep disturbance in CML patients treated with TKI therapy, which can have a debilitating impact on patients.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Diagnosis of CML on treatment with tyrosine kinase inhibitor.
3. On stable TKI therapy for at least 6 months duration
4. Confirmation of ongoing chronic phase
5. Male or females aged: 18 - 70 years old
6. On-going fatigue for more than 6 months with impairment in daily life activities/ or no fatigue as described in point 7.
7. If recruited to fatigue group then subjects would require both a - Chalder score > or = 5 and a Modified Fatigue Impact scale score > or = 43
8. If recruited to control group, then subjects would require both a Chalder score < or = 2 and a Modified Fatigue Impact Scale score <33

Exclusion Criteria:

1. Not currently on treatment with a TKI inhibitor.
2. Previous or active other neoplasm.
3. Past medical history including diagnosed sleep disorder, depression and on current therapy, sleep apnoea, uncontrolled thyroid dysfunction and neurological disorder
4. Active treatment with any of the following drug groups: anti cholinergic or anti muscarinic drugs, tricyclic antidepressants, serotonin norepinephrine reuptake inhibitors (SNRIs), selective serotonin reuptake inhibitors (SSRIs), Norepinephrine Dopamine Reuptake inhibitor (NDRI), Serotonin antagonist and reuptake inhibitor (SARI), Norepinephrine Antagonist serotonin antagonist (NASA), Monoamine oxidase inhibitors (MAO), regular sedating antihistamine use, regular opioid use, beta blockers, methyldopa, clonidine, benzodiazepines and zopiclone.
5. Prior allogeneic SCT
6. Have a history of alcohol or substance abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CML- Chronic phase patients in a single centre with significant fatigue on TKIs in group 1. In Group 2, CML chronic phase patients with no significant fatigue.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-05-12 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 14 days
  Assessed by validated questionnaires (Chalder and Modified Fatigue Impact scale), with scoring as described in eligibility criteria. Control group < or = 2 for Chalder score and < or = 33 for the MFIS score.For fatigue group a score > or = 5 for Chalder score and > or = 43 for the MFIS score.
Subjective sleep disturbance | 1 day
  Assessed by Pittsburgh Sleep Quality Index (validated). Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Subjective sleep | 14 days
  Assessed by sleep diary.
Percentage Sleep Efficiency | 14 days
  Percentage Sleep efficiency assessed using actigraphy accelerometer that can reliably translate physical motion and exerted energy into a numeric representation measured in 30 or 60-second epochs allowing continuous data collection over weeks. Percentage sleep efficiency is assessed, defined as the ratio between the total sleep time, and the total time dedicated to sleep (both sleeping and awake eg attempting to fall asleep or back asleep), measured in hours and minutes.
Sleep fragmentation index | 14 days
  Calculated by actigraphy using the total number of awakenings from deeper non-rapid eye movement to lighter sleep divided by the total sleep time in hours. Measured in hours and minutes.
Actigraphy variables | 14 days
  total sleep time (assumed sleep) measured using muscle motion/movement by accelerator in actigraphy monitor, and using algorithms that transform the raw accelerometer data into counts.
Actual wake time (wake after sleep onset) | 14 days
  Measured using accelerator in actigraphy monitor to assess objectively time to waking, measured in minutes and hours.

SECONDARY OUTCOMES:
Serum biomarker analysis | 1 day
  Activin B peripheral blood analysis, measured in pg/ml
Serum biomarker analysis | 1 day
  L-carnitine peripheral blood analysis, measured in umol/L

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Milojkovic, MbChB, PHD, Principal Investigator — Imperial NHS Healthcare Trust
Locations (1):
- Imperial NHS Healthcare Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data shared with coinvestigators will be anonymised.

REFERENCES:
- [Result] Innes AJ, Milojkovic D, Apperley JF. Allogeneic transplantation for CML in the TKI era: striking the right balance. Nat Rev Clin Oncol. 2016 Feb;13(2):79-91. doi: 10.1038/nrclinonc.2015.193. Epub 2015 Nov 17. PMID 26573423
- [Result] Efficace F, Baccarani M, Breccia M, Alimena G, Rosti G, Cottone F, Deliliers GL, Barate C, Rossi AR, Fioritoni G, Luciano L, Turri D, Martino B, Di Raimondo F, Dabusti M, Bergamaschi M, Leoni P, Simula MP, Levato L, Ulisciani S, Veneri D, Sica S, Rambaldi A, Vignetti M, Mandelli F; GIMEMA. Health-related quality of life in chronic myeloid leukemia patients receiving long-term therapy with imatinib compared with the general population. Blood. 2011 Oct 27;118(17):4554-60. doi: 10.1182/blood-2011-04-347575. Epub 2011 Jul 12. PMID 21750313
- [Result] Lidbury BA, Kita B, Lewis DP, Hayward S, Ludlow H, Hedger MP, de Kretser DM. Activin B is a novel biomarker for chronic fatigue syndrome/myalgic encephalomyelitis (CFS/ME) diagnosis: a cross sectional study. J Transl Med. 2017 Mar 16;15(1):60. doi: 10.1186/s12967-017-1161-4. PMID 28302133
- [Result] Cruciani RA, Zhang JJ, Manola J, Cella D, Ansari B, Fisch MJ. L-carnitine supplementation for the management of fatigue in patients with cancer: an eastern cooperative oncology group phase III, randomized, double-blind, placebo-controlled trial. J Clin Oncol. 2012 Nov 1;30(31):3864-9. doi: 10.1200/JCO.2011.40.2180. Epub 2012 Sep 17. PMID 22987089
- [Result] Bower H, Bjorkholm M, Dickman PW, Hoglund M, Lambert PC, Andersson TM. Life Expectancy of Patients With Chronic Myeloid Leukemia Approaches the Life Expectancy of the General Population. J Clin Oncol. 2016 Aug 20;34(24):2851-7. doi: 10.1200/JCO.2015.66.2866. Epub 2016 Jun 20. PMID 27325849
- [Result] Sadeh A. The role and validity of actigraphy in sleep medicine: an update. Sleep Med Rev. 2011 Aug;15(4):259-67. doi: 10.1016/j.smrv.2010.10.001. Epub 2011 Jan 14. PMID 21237680
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Sharf G, Marin C, Bradley JA, Pemberton-Whiteley Z, Bombaci F, Christensen RIO, Gouimi B, Deekes NB, Daban M, Geissler J. Treatment-free remission in chronic myeloid leukemia: the patient perspective and areas of unmet needs. Leukemia. 2020 Aug;34(8):2102-2112. doi: 10.1038/s41375-020-0867-0. Epub 2020 May 26. PMID 32457354
- [Result] Luik AI, Zuurbier LA, Hofman A, Van Someren EJ, Tiemeier H. Stability and fragmentation of the activity rhythm across the sleep-wake cycle: the importance of age, lifestyle, and mental health. Chronobiol Int. 2013 Dec;30(10):1223-30. doi: 10.3109/07420528.2013.813528. Epub 2013 Aug 23. PMID 23971909